CLINICAL TRIAL: NCT05785988
Title: Anti-Calcitonin Gene-Related Peptide (CGRP) Monoclonal Antibody Response After Switching in the Treatment of Migraine
Brief Title: Anti-CGRP Monoclonal Antibody Response After Switching (AMARAS)
Acronym: AMARAS
Status: Recruiting | Type: Observational
Sponsor: Hospital Clínico Universitario de Valladolid (Other)
Collaborators: Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León (Other)
Responsible Party: Principal Investigator, David García Azorín, Headache Unit, Department of Neurology, Principal Investigator, Hospital Clínico Universitario de Valladolid
Other Study IDs: PI-22-2658
Record Dates: First submitted 2023-03-11; First posted 2023-03-27 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Migraine; Head Pain
Keywords: Headache disorders; Painful disorders; Calcitonin gene-related peptide (CGRP)
MeSH Terms: conditions — Migraine Disorders; Headache; Headache Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with migraine treated with a second anti-CGRP: Patients with migraine treated with a second anti-CGRP monoclonal antibody as per responsible physician criteria in routine clinical practice.

SUMMARY:
Monoclonal antibodies targeting calcitonin gene-related peptide (mAb-CGRP) have shown efficacy and effectiveness in the treatment of episodic and chronic migraine, however, not all patients respond to them. Preliminary data suggests that some patients who failed to one of them, may respond to a different anti-CGRP monoclonal antibody.

Observational analytic study with a retrospective cohort design including patients treated with a second mAb-CGRP due to lack of response to the first one.

The aim of this study is to provide Class II evidence about the effectiveness and tolerability of the mAb-CGRP switching in patients with migraine, treated in a real-world setting.

DETAILED DESCRIPTION:
Background:

Migraine is the first cause of disability in the most active ages of life. Unlike other diseases, there are effective treatments that can lessen the burden of the disease. Currently, there are different treatments that act at different levels, many of them being non-migraine-specific and associated to poor tolerability. The monoclonal antibodies targeting calcitonin gene-related peptide (mAb-CGRP), or its receptor have shown efficacy in the treatment of episodic and chronic migraine, with a significantly lower rate of side effects. In Spain, the National Health System subsidizes them in patients with high-frequency episodic migraine or chronic migraine with prior failure to at least three preventive drugs.

There is preliminary evidence that suggest that approximately one-third of patients who have not responded to one mAb-CGRP may respond to a different mAb-CGRP, not necessarily with a different mechanism of action. The aim of this study is to provide Class II evidence about the effectiveness and tolerability of the mAb-CGRP switching in patients with migraine, treated in a real-world setting.

Study design:

Observational analytic study with a retrospective cohort design.

Endpoints:

The study endpoints will be based on the International Headache Society guidelines for controlled trials of chronic migraine, and will include effectiveness endpoints and safety endpoints.

Sample Size:

According to real-world data in our setting, the effectiveness rate of monoclonal antibodies in clinical practice conditions ranges between 40-60%. We aim to collect at least 300 patients treated with a secondary mAb-CGRP.

Methodology:

Observational analytic study with a retrospective cohort design. Spanish Hospitals with Headache Units or monographic headache consultations participate in the study. In all participant centers, patients carried out a headache diary that assesses the frequency of headache, migraine and acute treatment use.

Study intervention:

A structured questionnaire will be administered to patients, including demographic variables, such as sex, age at migraine onset, age at first mAb-CGRP use, age at second mAb-CGRP use. The following clinical variables were collected type of migraine (episodic / chronic), duration (in months) of high-frequency episodic migraine or chronic migraine; presence and type of aura; number and type of prior prophylactic drugs; mAb-CGRP used in first and second place; reason for discontinuation (lack of efficacy, lack of tolerability); frequency of headache, migraine, acute medication and triptan use per month; presence and type of adverse effects.

All the information was introduced in a standardize data collection form that will be hosted in RedCap.

Recruitment and sampling:

All consecutive patients treated with mAb-CGRP in the participating sites were screened for eligibility, including the administrative databases of all patients treated during the study period.

Data sources:

Paper or electronic health records was used, and structured headache diaries were provided to patients.

Ethics:

The study has been approved by the Ethics Review Board of East Valladolid (PI-22-2658). The study is conducted in accordance with the principles of the Declaration of Helsinki

Statistical Analysis:

First, a descriptive analysis will be carried out. The proportion of patients treated with a monoclonal antibody who receive treatment with a second will be described. A sub-group analysis will be done, depending on whether the reason for the mAb-CGRP switch an effectiveness failure or a tolerability failure was. The 50%, 30%, and 75% response rates will be calculated in the pre-specified study periods, as well as the frequency and type of adverse effects. To evaluate the reduction in days of headache per month, days of migraine, days of use of analgesics, and days of triptans, in the study periods, in relation to the baseline period, the Student's T-test for paired samples will be used. or the Mann-Whitney U, depending on the type of distribution of the sample. Normality of the sample will be assessed with the Kolmogorov-Smirnov test. To evaluate the predictors of response, a logistic regression analysis will be performed in which the independent variable will be the presence of a 50% response between weeks 8-12, and the rest of the study variables will be evaluated first by univariate regression, and after that, analysis multivariate in those with a P value less than 0.1.

Statistical analysis will be performed both by intention to treat (including all patients receiving treatment with a second monoclonal) and per-protocol analysis (those in which the information is complete). In case of missing data, for variables related to treatment, a conservative imputation will be performed using baseline-carried forward, for variables from 8-12 weeks and last-observation carried forward for variables from weeks 8-12.

A stratified analysis will be performed according to whether the reason for discontinuation of the first monoclonal antibody was the failure of effectiveness or lack of tolerance. A stratified analysis will also be performed in treatments between drugs directed against CGRP and their receptor A statistical significance level of 5% will be considered. The correction will be made for multiple comparisons by False Discovery Rate, using the Benjamini-Hochberg method.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age over 18 years old;
* 2. Confirmed diagnosis of migraine, according to the International Classification of Headche Disorders, 3rd version;
* 3. Treatment with a mAb-CGRP as per responsible physician criteria in routine clinical practice.

Exclusion Criteria:

* 1. Unavailability of information prior to the treatment use;
* 2. Other painful disorders that may interfere in the evaluation of the outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients treated with mAb-CGRP in the participating sites are screened for eligibility, including the administrative databases of all patients treated during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2024-11-10 (Estimated); Study Completion 2024-11-10 (Estimated)

PRIMARY OUTCOMES:
50% response weeks 8-12 | Between weeks 8-12 of treatment, compared to the month prior to the start of treatment
  To evaluate the proportion of patients with migraine treated with a second anti-CGRP monoclonal antibody that achieve a 50% response

SECONDARY OUTCOMES:
50% response weeks 20-24 | Between weeks 20-24 of treatment, compared to the month prior to the start of treatment
  To evaluate the proportion of patients with migraine treated with a second anti-CGRP monoclonal antibody that achieve a 50% response
50% response weeks 32-36 | Between weeks 32-36 of treatment, compared to the month prior to the start of treatment
  To evaluate the proportion of patients with migraine treated with a second anti-CGRP monoclonal antibody that achieve a 50% response
50% response weeks 44-48 | Between weeks 44-48 of treatment, compared to the month prior to the start of treatment
  To evaluate the proportion of patients with migraine treated with a second anti-CGRP monoclonal antibody that achieve a 50% response
30% response weeks 8-12 | Between weeks 8-12 of treatment, compared to the month prior to the start of treatment
  To evaluate the proportion of patients with migraine treated with a second anti-CGRP monoclonal antibody that achieve a 30% response
30% response weeks 20-24 | Between weeks 20-24 of treatment, compared to the month prior to the start of treatment
  To evaluate the proportion of patients with migraine treated with a second anti-CGRP monoclonal antibody that achieve a 30% response
30% response weeks 32-36 | Between weeks 32-36 of treatment, compared to the month prior to the start of treatment
  To evaluate the proportion of patients with migraine treated with a second anti-CGRP monoclonal antibody that achieve a 30% response
30% response weeks 44-48 | Between weeks 44-48 of treatment, compared to the month prior to the start of treatment
  To evaluate the proportion of patients with migraine treated with a second anti-CGRP monoclonal antibody that achieve a 30% response
75% response weeks 8-12 | Between weeks 8-12 of treatment, compared to the month prior to the start of treatment
  To evaluate the proportion of patients with migraine treated with a second anti-CGRP monoclonal antibody that achieve a 75% response
75% response weeks 20-24 | Between weeks 20-24 of treatment, compared to the month prior to the start of treatment
  To evaluate the proportion of patients with migraine treated with a second anti-CGRP monoclonal antibody that achieve a 75% response
75% response weeks 32-36 | Between weeks 32-36 of treatment, compared to the month prior to the start of treatment
  Evaluate the proportion of patients with migraine treated with a second anti-CGRP monoclonal antibody that achieve a 75% response
75% response weeks 44-48 | Between weeks 44-48 of treatment, compared to the month prior to the start of treatment
  To evaluate the proportion of patients with migraine treated with a second anti-CGRP monoclonal antibody that achieve a 75% response
Change in headache days per month weeks 8-12 | Between weeks 8-12 compared to the month prior to starting treatment
  To evaluate the change in headache days per month
Change in migraine days per month weeks 8-12 | Between weeks 8-12 compared to the month prior to starting treatment
  To evaluate the change in migraine days per month
Change in days of use of symptomatic medication per month weeks 8-12 | Between weeks 8-12 with respect to the month prior to the start of treatment
  To evaluate the change in days of use of symptomatic medication per month
Change in days of use of triptan per month weeks 8-12 | Between weeks 8-12 with respect to the month prior to the start of treatment
  To evaluate the change in days of triptan use per month
Change in headache days per month weeks 20-24 | Between weeks 20-24 compared to the month prior to starting treatment
  To evaluate the change in headache days per month
Change in migraine days per month weeks 20-24 | Between weeks 20-24 compared to the month prior to starting treatment
  To evaluate the change in migraine days per month
Change in days of use of symptomatic medication per month weeks 20-24 | Between weeks 20-24 with respect to the month prior to the start of treatment
  To evaluate the change in days of use of symptomatic medication per month
Change in days of use of triptan per month weeks 20-24 | Between weeks 20-24 with respect to the month prior to the start of treatment
  To evaluate the change in days of use of triptans per month
Change in headache days per month weeks 32-36 | Between weeks 32-36 compared to the month prior to starting treatment
  To evaluate the change in headache days per month
Change in migraine days per month weeks 32-36 | Between weeks 32-36 compared to the month prior to starting treatment
  To evaluate the change in migraine days per month
Change in days of use of symptomatic medication per month weeks 32-36 | Between weeks 32-36 with respect to the month prior to the start of treatment
  To evaluate the change in days of use of symptomatic medication per month
Change in days of use of triptan per month weeks 32-36 | Between weeks 32-36 compared to the month prior to the start of treatment
  To evaluate the change in days of triptan use per month
Change in headache days per month weeks 44-48 | Between weeks 44-48 compared to the month prior to starting treatment
  To evaluate the change in headache days per month
Change in migraine days per month weeks 44-48 | Between weeks 44-48 compared to the month prior to starting treatment
  To evaluate the change in migraine days per month
Change in days of use of symptomatic medication per month weeks 44-48 | Between weeks 44-48 with respect to the month prior to the start of treatment
  To evaluate the change in days of use of symptomatic medication per month
Change in days of use of triptan per month weeks 44-48 | Between weeks 44-48 compared to the month prior to starting treatment
  To evaluate the change in days of triptan use per month
Frequency and type of adverse events | Through study completion, an average of 1 year
  To assess the frequency and type of treatment-related adverse events
Adverse events leading to treatment discontinuation | Through study completion, an average of 1 year
  To evaluate the proportion of patients who discontinue treatment due to an adverse effect
Predictors of 50% response | Between weeks 8-12, in relation to the month prior to the start of treatment
  To explore possible predictors of response, using as a response variable the presence of a 50% response

CONTACTS AND LOCATIONS:
Overall Officials: David García Azorín, MD, PhD, Principal Investigator — Research coordinator
Locations (1):
- Hospital Clínico Universitario de Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data may be shared upon reasonable request to the principal investigator.

REFERENCES:
- [Background] Steiner TJ, Stovner LJ, Jensen R, Uluduz D, Katsarava Z; Lifting The Burden: the Global Campaign against Headache. Migraine remains second among the world's causes of disability, and first among young women: findings from GBD2019. J Headache Pain. 2020 Dec 2;21(1):137. doi: 10.1186/s10194-020-01208-0. No abstract available. PMID 33267788
- [Background] Deuschl G, Beghi E, Fazekas F, Varga T, Christoforidi KA, Sipido E, Bassetti CL, Vos T, Feigin VL. The burden of neurological diseases in Europe: an analysis for the Global Burden of Disease Study 2017. Lancet Public Health. 2020 Oct;5(10):e551-e567. doi: 10.1016/S2468-2667(20)30190-0. PMID 33007212
- [Background] GBD 2016 Neurology Collaborators. Global, regional, and national burden of neurological disorders, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2019 May;18(5):459-480. doi: 10.1016/S1474-4422(18)30499-X. Epub 2019 Mar 14. PMID 30879893
- [Background] Charles A. The pathophysiology of migraine: implications for clinical management. Lancet Neurol. 2018 Feb;17(2):174-182. doi: 10.1016/S1474-4422(17)30435-0. Epub 2017 Dec 8. PMID 29229375
- [Background] Ashina M, Terwindt GM, Al-Karagholi MA, de Boer I, Lee MJ, Hay DL, Schulte LH, Hadjikhani N, Sinclair AJ, Ashina H, Schwedt TJ, Goadsby PJ. Migraine: disease characterisation, biomarkers, and precision medicine. Lancet. 2021 Apr 17;397(10283):1496-1504. doi: 10.1016/S0140-6736(20)32162-0. Epub 2021 Mar 25. PMID 33773610
- [Background] Charles A, Pozo-Rosich P. Targeting calcitonin gene-related peptide: a new era in migraine therapy. Lancet. 2019 Nov 9;394(10210):1765-1774. doi: 10.1016/S0140-6736(19)32504-8. Epub 2019 Oct 23. PMID 31668411
- [Background] Drellia K, Kokoti L, Deligianni CI, Papadopoulos D, Mitsikostas DD. Anti-CGRP monoclonal antibodies for migraine prevention: A systematic review and likelihood to help or harm analysis. Cephalalgia. 2021 Jun;41(7):851-864. doi: 10.1177/0333102421989601. Epub 2021 Feb 10. PMID 33567891
- [Background] Gantenbein AR, Agosti R, Gobbi C, Flugel D, Schankin CJ, Viceic D, Zecca C, Pohl H. Impact on monthly migraine days of discontinuing anti-CGRP antibodies after one year of treatment - a real-life cohort study. Cephalalgia. 2021 Oct;41(11-12):1181-1186. doi: 10.1177/03331024211014616. Epub 2021 May 17. PMID 34000847
- [Background] Vernieri F, Altamura C, Brunelli N, Costa CM, Aurilia C, Egeo G, Fofi L, Favoni V, Pierangeli G, Lovati C, Aguggia M, d'Onofrio F, Doretti A, Di Fiore P, Finocchi C, Rao R, Bono F, Ranieri A, Albanese M, Cevoli S, Barbanti P; GARLIT Study Group. Galcanezumab for the prevention of high frequency episodic and chronic migraine in real life in Italy: a multicenter prospective cohort study (the GARLIT study). J Headache Pain. 2021 May 3;22(1):35. doi: 10.1186/s10194-021-01247-1. PMID 33941080
- [Background] Overeem LH, Peikert A, Hofacker MD, Kamm K, Ruscheweyh R, Gendolla A, Raffaelli B, Reuter U, Neeb L. Effect of antibody switch in non-responders to a CGRP receptor antibody treatment in migraine: A multi-center retrospective cohort study. Cephalalgia. 2022 Apr;42(4-5):291-301. doi: 10.1177/03331024211048765. Epub 2021 Oct 13. PMID 34644203
- [Background] Porta-Etessam J, Gonzalez-Garcia N, Guerrero AL, Garcia-Azorin D. Failure to monoclonal antibodies against CGRP or its receptor does not preclude lack of efficacy to other drugs from the same therapeutic class. Neurologia (Engl Ed). 2020 Nov 8:S0213-4853(20)30312-1. doi: 10.1016/j.nrl.2020.10.009. Online ahead of print. No abstract available. English, Spanish. PMID 33176918
- [Background] Ferreira JA. The Benjamini-Hochberg method in the case of discrete test statistics. Int J Biostat. 2007;3(1):Article 11. doi: 10.2202/1557-4679.1065. PMID 22550651